CLINICAL TRIAL: NCT05397886
Title: Comparison of Remimazolam With Flumazenil vs. Propofol TIVA During RFCA for Atrial Fibrillation
Brief Title: Comparison of Remimazolam With Flumazenil vs. Propofol During RFCA for Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Yunseok Jeon, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Remimazolam_RFCA
Record Dates: First submitted 2022-05-09; First posted 2022-05-31 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Recovery
Keywords: recovery; remimazolam; flumazenil; propofol; radiofrequency catheter ablation
MeSH Terms: interventions — Flumazenil; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remimazolam with flumazenil (Experimental): Patients allocated to remimazolam with flumazenil group receives remimazolam as the main anesthetics during general anesthesia and then flumazenil administration at the end of anesthesia. Remifentanil continuous infusion can be used for hemodynamic stability and analgesia.
  Interventions: Drug: Remimazolam Besylate; Drug: Flumazenil
- Propofol total intravenous anesthesia (Active Comparator): Patients allocated to propofol total intravenous anesthesia group receives propofol as the main anesthetics during general anesthesia until the end of anesthesia. Remifentanil continuous infusion can be used for hemodynamic stability and analgesia.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Remimazolam Besylate — Remimazolam Besylate is used as intervention drug for general anesthesia, which followed by flumazenil administration at the end of anesthesia, to be compared to propofol total intravenous anesthesia during radiofrequency catheter ablation of atrial fibrillation.
  Arms: Remimazolam with flumazenil
Drug: Flumazenil — Flumazenil is used as additional intervention drug to facilitate emergence from general anesthesia in the Remimazolam with Flumazenil group.
  Arms: Remimazolam with flumazenil
Drug: Propofol — Propofol is used as active comparator drug for general anesthesia until the end of anesthesia, to be compared to remimazolam besylate during radiofrequency catheter ablation of atrial fibrillation.
  Arms: Propofol total intravenous anesthesia

SUMMARY:
This prospective randomized trial aims to compare recovery time from discontinuation of remimazolam followed by flumazenil administration vs. propofol total intravenous anesthesia as the main general anesthetics during radiofrequency catheter ablation treatment of atrial fibrillation.

DETAILED DESCRIPTION:
Adult patients with atrial fibrillation undergoing radiofrequency catheter ablation under general anesthesia are randomized to receive either remimazolam with flumazenil or propofol total intravenous anesthesia as the main anesthetics. After completion of radiofrequency ablation, each anesthetic is discontinued. The primary outcome of the study is comparison of the time to the first eye opening responding to doctor's command from the discontinuation of each drug between the groups. Secondary outcomes includes the time to removal of supraglottic laryngeal mask airway device from discontinuation of each drug, incidence of three consecutive hypotension (systolic blood pressure under 80 mmHg) recordings at 2.5 min-intervals, and intraprocedural vasoactive-inotropic score.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient, age 20-75 years, scheduled for radiofrequency catheter ablation of atrial fibrillation under general anesthesia

Exclusion Criteria:

* Patients who are not alert before procedure
* Hemodynamicaly unstable patients before procedure
* Patients with history of adverse reaction of allergic reaction to study drugs
* Patients who are anticipated to be unable to remove supraglottic airway or endotracheal tube due to severe dyspnea or need for mechanical ventilatory support
* Use of sedatives (anxiolytics, psychoactive medication, antidepressants, hypnotics) within 24 h
* Known galactose intolerance, Lapp lactase deficiency, glucose-galactose malabsorption
* Severe hepatic or renal dysfunction
* Alcohol or drug dependence
* Organic brain disorder
* Spinal or cerebellar ataxia
* Acute narrow-angle glaucoma
* Patients with shock or coma
* Pregnant or lactating women
* Patients with hypersensitive to beans or peanut
* Patients who refuse to participate

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2022-08-02 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2023-04-25 (Actual)

PRIMARY OUTCOMES:
Time to eye opening | up to 1 hour
  Time to first eye opening responding to doctor's command from discontinuation of main anesthetics

SECONDARY OUTCOMES:
Time to remove laryngeal mask airway | up to 1 hour
  Time to removal of supraglottic laryngeal mask airway from discontinuation of main anesthetics
Incidence of hypotension | During anesthesia for radiofrequency ablation procedure
  Incidence of three consecutive hypotension, which is defined as systolic blood pressure under 80 mmHg, at 2.5 min-intervals
Vasoactive-inotropic score | During anesthesia for radiofrequency ablation procedure
  Intraprocedural vasoactive-inotropic score, which is calculated as: dopamine dose (μg/kg/min) + dobutamine dose (μg/kg/min) + 100 х epinephrine (μg/kg/min) + 100 х norepinephrine (μg/kg/min) + 10000 х vasopressin (unit/kg/min)

CONTACTS AND LOCATIONS:
Overall Officials: Yunseok Jeon, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lee S, Lee J, Hwang SY, Ju JW, Nam K, Ahn HJ, Lee SR, Choi EK, Jeon Y, Cho YJ. Remimazolam-flumazenil provides fast recovery from general anesthesia compared to propofol during radiofrequency catheter ablation of atrial fibrillation. Sci Rep. 2024 Jun 3;14(1):12660. doi: 10.1038/s41598-024-63578-8. PMID 38831029